CLINICAL TRIAL: NCT00341107
Title: Physicians Survey on Genetic Testing
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999999010; OH99-C-N010
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2006-01

CONDITIONS: Cancer
Keywords: Cancer; Genes; Screening; Primary Care; Inherited Susceptibility
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease

SUMMARY:
Research and development in genetic testing for cancer susceptibility genes has advanced rapidly in recent years, allowing healthy individuals, cancer patients, and their families to determine if they carry mutations which increase their risk of breast, ovarian, prostate, colon, and other cancers. Initial efforts have unfolded primarily in academic medical centers targeting families at high risk for cancer. There is currently no information available for assessing the prevalence of genetic testing for cancer susceptibility genes at the national level, or for evaluating the knowledge of and attitudes toward such testing among primary care physicians. The objectives of this survey are to determine the utilization of genetic tests by physicians at the national level; to ascertain physician knowledge of available genetic tests for specific cancer susceptibility genes, to examine physicians' general attitudes toward testing, and; to explore possible variation in utilization and knowledge/attitudes by medical specialty, type of practice, year of training completion, board status, urbanicity, and geographic region. The primary research question that this survey will address is what is the prevalence of use of genetic testing for cancer susceptibility among primary care physicians in the U.S.? The survey will also assess whether there are statistically significant differences in 1) self-reported knowledge, current use of, and future intentions to use genetic testing for cancer susceptibility, and 2) perceptions of barriers to testing, among primary care physicians by their type and location of practice, and recency of training. Primary care physicians (internists, obstetrician/gynecologist, family and general practitioners) will also be compared with specialty groups (gastroenterologists, surgeons, urologists) and oncologists with respect to their use, attitudes towards, and knowledge of, genetic testing for cancer susceptibility. A questionnaire is being administered by mail, telephone, facsimilie or Internet to a nationally representative sample of 2,100 physicians. Responding physicians select their preferred response mode. Study participants are primary care and specialty physicians with active licenses to practice medicine in the U.S. A data file with personal identifiers deleted will be prepared for statistical analysis to estimate the prevalence and determine predictors of use and intentions to genetic tests for inherited cancer susceptibility.

DETAILED DESCRIPTION:
Research and development in genetic testing for cancer susceptibility genes has advanced rapidly in recent years, allowing healthy individuals, cancer patients, and their families to determine if they carry mutations which increase their risk of breast, ovarian, prostate, colon, and other cancers. Initial efforts have unfolded primarily in academic medical centers targeting families at high risk for cancer. There is currently no information available for assessing the prevalence of genetic testing for cancer susceptibility genes at the national level, or for evaluating the knowledge of and attitudes toward such testing among primary care physicians. The objectives of this survey are to determine the utilization of genetic tests by physicians at the national level; to ascertain physician knowledge of available genetic tests for specific cancer susceptibility genes, to examine physicians' general attitudes toward testing, and; to explore possible variation in utilization and knowledge/attitudes by medical specialty, type of practice, year of training completion, board status, urbanicity, and geographic region. The primary research question that this survey will address is what is the prevalence of use of genetic testing for cancer susceptibility among primary care physicians in the U.S.? The survey will also assess whether there are statistically significant differences in 1) self-reported knowledge, current use of, and future intentions to use genetic testing for cancer susceptibility, and 2) perceptions of barriers to testing, among primary care physicians by their type and location of practice, and recency of training. Primary care physicians (general internists, obstetrician/gynecologist, family and general practitioners) will also be compared with specialty groups (gastroenterologists, surgeons, urologists) and oncologists with respect to their use, attitudes towards, and knowledge of, genetic testing for cancer susceptibility. A questionnaire was administered by mail, telephone, facsimilie or Internet to a nationally representative sample of 1,251 primary care physicians and specialists. Study participants are primary care and specialty physicians with active licenses to practice medicine in the U.S. A data file with personal identifiers deleted will be prepared for statistical analysis to estimate the prevalence and determine predictors of use and intentions to genetic tests for inherited cancer susceptibility.

ELIGIBILITY:
* INCLUSION CRITERIA:

All physicians in the U.S. commonly considered to be adult primary care practitioners: family practitioners, general practitioners, general internists, and obstretrician/gynecologists (excluding physicians who practice only obstetrics).

For comparison purposes, physicians in the specialties of oncology, general surgery, gastroenterology and urology will also be included since they treat cancer patients and individuals at high risk for cancer.

EXCLUSION CRITERIA:

Physicians who are retired and/or do not hold active licenses, involved in full-time teaching, research or administration and not clinical practice, and physicians in training who are not yet board-eligible for their specialty re excluded from selection for the survey.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1350
Dates: Start 1999-02